CLINICAL TRIAL: NCT04539912
Title: Comparison of the Short-term Clinical Efficacy of Angulated Screw-retained and Cemented Single Implant Crowns in Esthetic Region: A Randomized Controlled Clinical Trial
Brief Title: Clinical Efficacy of Angulated Screw-retained and Cemented Single Implant Crowns in Esthetic Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Junyu Shi (Other)
Responsible Party: Sponsor-Investigator, Junyu Shi, Principal Investigator, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Organization: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: sh9th-20-09
Record Dates: First submitted 2020-09-01; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Angulated Screw-retained; Esthetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- angulated screw-retained group(AG) (Experimental)
  Interventions: Device: angulated screw retained crown
- cemented group (CG) (Active Comparator)
  Interventions: Device: cemented crown

INTERVENTIONS:
Device: angulated screw retained crown — ASC abutment was used in AG;
  Arms: angulated screw-retained group(AG)
Device: cemented crown — prefabricated Ti abutment was used in CG
  Arms: cemented group (CG)

SUMMARY:
Objective: To compare the clinical efficacy of angulated screw-retained and cemented single implant crowns(SIC) in esthetic region.

Methods/Design: The study was a prospective, single center, randomized controlled clinical trial. Patients with the needs of single tooth restoration in esthetics region were recruited from Oct. 2018 to Aug. 2019. Sixty patients were enrolled in the present study and they were randomly assigned into two groups: angulated screw-retained group(AG, 30 patients) and cemented group (CG,30 patients). Clinical and radiological evaluations were performed on the day of final crowns delivery and 12 months later. Implant survival rate, marginal bone loss(MBL), pro-inflammatory cytokinesin peri-implant crevicular fluid (PICF)(TNF-α, IL-6), mechanical complications, peri-implant conditions(mPI, PD, BOP%), pink esthetics score/white esthetics score (PES/ WES) and patients satisfaction were assessed.

ELIGIBILITY:
Inclusion Criteria:

* 1) age≥18;
* 2) Single dental implant in the esthetic region;
* 3) adjacent to natural teeth;
* 4) absence of oral mucosal disease and oral infection;
* 5)implants withconical connection (Nobel Active, Nobel Biocare® or NobelReplace Conical Connection, Nobel Biocare®);
* 6)patients with the willingness of all-ceramic permanent restorations.

Exclusion Criteria:

* 1)Multiple implants in the esthetic region, or the restoration is a bridge;
* 2)Heavy smokers (>10 cigarettes/day);
* 3) the angle between implant axis and restoration axis>25°;
* 4) uncontrolled periodontitis;
* 5) with systematic diseases that may affect implant therapy, such as uncontrolled diabetes mellitus (Fasting blood-glucose>7.2mmol/L, Glycosylated hemoglobin >7%), current intake of bisphosphonates (treatment for malignancy), pregnant(or plan to get pregnant), with history of radiation therapy in head and neck region;
* 6) Unwilling to participate in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Marginal bone loss | 1year
  Peri-apical radiographs with paralleling technique wereperformed on the day offinal restorations delivery and 1-year visit. Implant length was used as calibration reference. The distance between restoration margin and the most coronal level of implant-bone contactwas recorded. Final result was calculated as themean value of the mesial and distal sites

SECONDARY OUTCOMES:
Survival rate. | 1 year
  Survival rates were defined as the percentage of success implants and remained crowns which never been replaced
Pro-inflammatory cytokinesin peri-implant crevicular fluid (PICF) | 1 year
  we collected the patients' PICF with the paper strip (PerioPaper Strips; Oraflow Inc., Smithtown, NY, USA) at 1year follow-up to access differences in pro-inflammatory cytokines (IL-6 and TNF-α) between two groups.
Mechanical complications | 1 year
  Abutments or implants fracture and screw loosening or fracture
pocket probing depth(PD) | 1 year
  The depth of 6 sites（mesial, middle and distal of buccal/lingual ） was measured and the average value was calculated.
PES/WES | 1 year
  specific dentists were asked to give scores for variables of PES (Mesial papilla, distal papilla, level of soft-tissue margin, soft-tissue contour, alveolar process and soft-tissue color and texture) and WES (Tooth form, tooth volume/outline, color, surface texture and transparency) with the 2-1-0 scoring system. Final PES/WES was the sum the two. Total scores were defined as perfect rate (PES/WES≥22), acceptable rate (22>PES/WES≥15) and unfavorable rate (PES/WES<15).
Patient's satisfaction | 1 year
  patient's satisfaction(PS) with aesthetics, function and comfort of the restoration at 1-year visit. 0 score was extremely dissatisfied and 10 score was extremely satisfied. We also defined the final scores as perfect rate(PS≥9), acceptable rate(9>PS≥6) and unfavorable rate (PS<6).
bleeding on probing% (BOP%) | 1 year
  The BOP of 6 sites（mesial, middle and distal of buccal/lingual ） was probed and the percentage of BOP(+) was calculated.
modified plaque index (mPI) | 1 year
  Score 0; No detection of plaque Score 1: Plaque only recognized by running a probe across the smooth marginal surface of the implant. Implants covered by titanium spray in this area always score 1.
  Score 2: Plaque can be seen by the naked eye. Score 3: Abundance of soft matter.

CONTACTS AND LOCATIONS:
Locations (1):
- Jun-Yu Shi, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided